CLINICAL TRIAL: NCT05928169
Title: Determinants of Chronic Inflammatory Skin Disease Trajectories
Status: Recruiting | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Prof. Dr. Stephan Weidinger, Prof. Dr. Stephan Weidinger, University Hospital Schleswig-Holstein
Other Study IDs: D452/23
Record Dates: First submitted 2023-06-01; First posted 2023-07-03 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Atopic Dermatitis; Psoriasis; Lichen Planus; Alopecia Areata; Hidradenitis Suppurativa; Prurigo Nodularis; Cutaneous Lupus; Rosacea
Keywords: Inflammatory Skin Diseases
MeSH Terms: conditions — Dermatitis, Atopic; Psoriasis; Lichen Planus; Alopecia Areata; Hidradenitis Suppurativa; Rosacea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Skin biopsies, skin tape strips, skin swabs, blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Topical and systemic drugs — Recruitment and follow-up will be independent on the type of treatment

SUMMARY:
Although it is well known that the clinical expression and course of chronic inflammatory skin diseases are highly variable, there are insufficient epidemiological data on this, and the factors that determine the manifestation, clinical features and course are also largely unknown. There are currently no reliable markers that could predict or delineate patient subgroups to support patient management. The aim of this project is to identify clinical and molecular factors that correlate with disease, disease subtypes and progression through in-depth long-term clinical characterization of patients with chronic inflammatory skin diseases and examination of individual biomaterials.

DETAILED DESCRIPTION:
Chronic inflammatory skin diseases such as atopic dermatitis (AD), psoriasis (Pso) and Hidradenitis suppurativa (HS) are very heterogeneous diseases. Onset, clinical features, disease severity, individual trigger factors and response to therapy vary widely between patients and over time, presenting a clinical challenge for diagnosis, counseling, and individualization of management. With the growing interest in inflammatory skin diseases, the need has been recognized to better investigate their natural course and trajectories, associations with environmental and lifestyle factors, and clinical and molecular features underlying their heterogeneity. Initial pilot studies suggested disease subtypes that differ molecularly and/or clinically; however, molecular profiles in particular are subject to variation over time and not necessarily stable. To confirm and extend such preliminary observations, a larger cohort of patients will be studied with careful longitudinal clinical characterization as well as repeatedly obtained specimens, in order to gain deeper insights into disease dynamics. In particular, we will search for clinical and molecular factors that correlate with disease progression and subtypes, and investigate variability in the regulation of molecular mechanisms over time and at resolution and flare-ups.

ELIGIBILITY:
Inclusion Criteria:

* dermatologist-diagnosed inflammatory skin disease
* informed consent

Exclusion Criteria:

* subject and/or the legal guardians are not able to give written informed consent
* pregnant and breastfeeding women
* concurrent participation in a clinical trial
* use of systemic immunosuppressive therapy or phototherapy during the last 4 weeks or receipt of biologics therapy (e.g. dupilumab, tralokinumab) within the last 3 months
* treatment of the target skin areas with topical corticosteroids, calcineurin inhibitors or emollients 24 hours before sample collection

Ages: 0 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic inflammatory skin disease Healthy control individuals
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2032-04-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Physician-assessed global disease activity | Baseline, week 2, week 4, every 3 months up to 2 years
  Change in Investigator Global Assessment (IGA, 0-5)
Patient-reported global disease activity | Baseline, week 2, week 4, every 3 months up to 2 years
  Change in Patient Global Assessment (IGA, 0-5)

SECONDARY OUTCOMES:
Molecular features | Baseline, week 2, week 4, every 3 months up to 2 years
  Molecular and histopathological profiles in lesional skin and blood compared across diseases, over time and in response to therapy

CONTACTS AND LOCATIONS:
Overall Officials: Sascha Gerdes, MD, Study Director — University Hospital Schleswig-Holstein
Locations (1):
- Department of Dermatology and Allergy, University Hospital Schleswig-Holstein, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No
IPD can be made available only to individual collaborating researchers in compliance with other researchers in line with national as well as international data protection laws (e.g. GDPR, DSGVO)